CLINICAL TRIAL: NCT05737680
Title: Efficacy and Safety of Hydroxychloroquine in Colchicine-RESistant Glucocorticoid-DependenT IdiOpathic REcurrent Pericarditis: A Randomized Clinical Trial (The RESTORE Randomized Clinical Trial)
Brief Title: Hydroxychloroquine in Colchicine-Resistant Glucocorticoid-Dependent Idiopathic Recurrent Pericarditis
Acronym: RESTORE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Prof. Konstantinos P. Tsioufis, MD, PhD, FESC, FACC, Professor of Cardiology, Director of 1st Department of Cardiology, Hippokratio Hospital, University of Athens, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RESTORE
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Pericarditis Idiopathic Recurrent
MeSH Terms: interventions — Hydroxychloroquine; Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine arm (Active Comparator): Hydroxychloroquine 400mg daily
  Interventions: Drug: Hydroxychloroquine
- Colchicine arm (Active Comparator): Colchicine continued
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 400mg daily
  Arms: Hydroxychloroquine arm
Drug: Colchicine — Colchicine continued
  Arms: Colchicine arm

SUMMARY:
Among patients with colchicine-resistant glucocorticoid-dependent idiopathic RP (idiopathic recurrent pericarditis during at least a second recurrence, having met the 2015 European Society of Cardiology criteria for pericarditis at least once), HCQ 400mg daily is associated with a reduce the risk of recurrence.

The above hypothesis will be tested with a randomized, prospective, parallel, open label clinical trial. The expected study duration is approximately 12 months from the time the first subject is enrolled (planned for February 2023) to the time of study's termination date (December 2024). The researchers will obtain approval by the institutional review board (IRB).

DETAILED DESCRIPTION:
Recurrent pericarditis (RP) along with pericardial tamponade and constrictive pericarditis are potential complications of acute pericarditis. They appear most frequently in secondary forms of pericarditis as compared with idiopathic acute pericarditis. Among the above-mentioned complications, RP is a highly problematic and disabling condition, which severely impairs the quality of life of affected patients, since it often requires emergency department visits and hospitalizations.

Moreover, the side effects of treatment constitute an additional concern both for the managing physicians and affected patients. In the most recent guidelines for the diagnosis and management of pericardial diseases of the European Society of Cardiology (ESC), a stepwise approach has been proposed for the treatment of RP including 4 treatment lines according to disease severity and individual response to treatment. Among them hydroxychloroquine (HCQ), an anti-malarial drug with immunomodulatory properties could potentially have a role as a third step treatment. HCQ, is an established treatment for all patients with systemic lupus erythematosus (SLE) including those with serositis (pericarditis, pleuritis) but data on HCQ efficacy for refractory idiopathic RP (IRP) are very scant.

The potential Anti-interleukin-1 agents are characterized by some disadvantages such as a long duration of therapy as well as high costs. In addition to this, only patients with a clear inflammatory pattern are candidates. Patients with mild or doubtful symptoms and/or normal or near normal levels of C-Reactive protein are not good candidates for anti-IL-1 therapy.

The investigators propose a randomized, prospective, parallel, open label, clinical trial, which will provide data on the efficacy and safety of HCQ in colchicine-resistant glucocorticoid-dependent idiopathic RP. The trial will have two study arms: HCQ 400mg daily vs. Colchicine continued. Patients with RP (idiopathic recurrent pericarditis during at least a second recurrence, having met the 2015 European Society of Cardiology criteria for pericarditis at least once) will be randomized to HCQ vs. Colchicine and will receive optimal post-recurrence care (increase the dose of methylprednisolone by 8 mg and then decrease by 2 mg every 2 weeks) in both arms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged≥18 years
* Idiopathic recurrent pericarditis with at least 2 recurrences
* Recurrent pericarditis defined as a first episode of acute pericarditis followed by recurrences (at least two recurrences for this study). First episode of pericarditis is diagnosed when at least two of the following criteria were present: pericarditis typical chest pain (sharp and pleuritic, improved by sitting up and leaning forward), pericardial friction rubs, widespread ST segment elevation or PR interval (PR) depressions not previously reported, and new or worsening pericardial effusion. Recurrence is diagnosed when chest pain recurs and one or more of the following signs is present: fever, pericardial friction rub, ECG changes, echocardiographic evidence of new or worsening pericardial effusion, and elevations in the white blood cell count, erythrocyte sedimentation rate or C-reactive protein. To be enrolled in this study, elevation of C-reactive protein is mandatory both in the first attack and in the following recurrences. The investigators differentiate recurrences from incessant pericarditis, term used to define patients with continued activity of pericarditis (with a symptom-free interval of < 6 weeks)
* Specific aetiologies excluded, including tuberculous, neoplastic or purulent aetiologies, post-cardiac injury syndromes, and rheumatic autoimmune diseases.
* Female subjects must be postmenopausal, or incapable of pregnancy or permanently sterile, or if of childbearing potential must agree to use highly-effective method of contraception.
* Signed written informed consent by the patient for participation in the study and agreement to comply with the medication and the follow-up schedule.

Exclusion Criteria:

* Ophthalmologic contraindications
* Structural heart disease
* Corrected QT interval >440msec in men and >450msec in women
* Left ventricular hypertrophy >13mm in men and >11mm in woman
* Known allergy or intolerance to hydroxychloroquine
* Life expectancy of < 12 months
* Complex congenital heart disease
* History of ventricular arrhythmias other than isolated extrasystoles
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal)
* Known channelopathy such as Brugada syndrome, long QT syndrome, or Catecholaminergic monomorphic ventricular tachycardia
* On the heart transplant list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate | 12 months follow-up
  The diagnosis of RP in a patient with history of a documented episode of acute pericarditis according to ESC guidelines was established in the presence of at least 2 of the following conditions: i. pleuritic chest pain, ii. pericardial friction rub, iii. ECG compatible with acute pericarditis and iv. first detected or increasing in size pericardial effusion. C-reactive protein (CRP) elevation was considered a confirmatory finding. Since RP frequently underlines a secondary etiology, an extensive work-up was performed to exclude such diseases. In particular, apart from the first line evaluation, second level investigations were additionally performed such as thyroid function tests, chest and abdominal computed tomography, serological screening for autoimmune disorders, serum tumor markers and QuantiFERON-Tuberculosis Gold test.

SECONDARY OUTCOMES:
Time to Pericarditis Recurrence | 12 months follow-up
  Time to pericarditis recurrence (from randomization to 1st recurrence). Kaplan-Meier. Clinical Events Committee (CEC)-confirmed recurrences used for primary analysis.
Dose of the Corticosteroid in the time of the recurrence | 12 months follow-up
State-Trait Anxiety Inventory (STAI) | 3,6,9,12 months follow-up
  This score measures two types of anxiety- state anxiety (S-anxiety) and trait anxiety (T-anxiety). It includes 40 self-reported items on a 4-point Likert scale. The scores range from 20 to 80, with higher scores correlating with greater anxiety. The 4-point scale for S-anxiety is as follows: 1) not at all, 2) somewhat, 3.) moderately so, 4) very much so. The 4-point scale for T-anxiety is as follows: 1) almost never, 2) sometimes, 3) often, 4) almost always.
Change over time of pericardial pain | 3,6,9,12 months follow-up
  Quantified using the four-point pain verbal rating scale (VRS-4). Minimum: 0, maximum: 3). Higher score indicates worse outcomes.
Change over time of C-reactive protein levels | 3,6,9,12 months follow-up
  Measured in mg/dL
Change over time of echocardiographic effusion | 3,6,9,12 months follow-up
  Measured in ml
Incidence and severity of Adverse Events | 3,6,9,12 months follow-up
  All adverse events (AEs) will be monitored and recorded to assess the tolerability and safety of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- "Hippokration" General Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided